CLINICAL TRIAL: NCT05019755
Title: A Randomized, Open-label, Single-dose, 2-way Crossover Clinical Trial to Investigate the Effect of Food on the Pharmacokinetics of IN-A002 Capsule in Healthy Male Subjects
Brief Title: A Study to Investigate the Effect of Food on the Pharmacokinetics of IN-A002 Capsule in Healthy Male Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IN_JSI_103
Record Dates: First submitted 2021-08-09; First posted 2021-08-25 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Healthy
MeSH Terms: interventions — Capsules

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A(First period) to B(Second period) order (Experimental): A: Oral Administration of IN-A002(IN-115314) in fasting status
  B: Oral Administration of IN-A002(IN-115314), 30 minutes after high-fat diet
  There will be a wash out period of 7days between period
  Interventions: Drug: IN-A002(IN-115314) capsule
- B(First period) to A(Second period) order (Experimental): B: Oral Administration of IN-A002(IN-115314), 30 minutes after high-fat diet
  A: Oral Administration of IN-A002(IN-115314) in fasting status
  There will be a wash out period of 7days between period
  Interventions: Drug: IN-A002(IN-115314) capsule

INTERVENTIONS:
Drug: IN-A002(IN-115314) capsule — Oral Administration of IN-A002(IN-115314), single dose
  Arms: A(First period) to B(Second period) order
Drug: IN-A002(IN-115314) capsule — Oral Administration of IN-A002(IN-115314), single dose
  Arms: B(First period) to A(Second period) order

SUMMARY:
This study aims to investigate the effect of food on the pharmacokinetics of IN-A002 capsule in healthy male subjects

DETAILED DESCRIPTION:
To explore the effect of High-fat diet on the pharmacokinetics of single dose of IN-A002 capsule in healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy male adults aged 19 to 55 years (inclusive) at the time of signing the informed consent form.
* Body mass index (BMI) ≥ 18.0 and ≤ 30.0 kg/m^2 with a body weight ≥ 50.0 kg and ≤ 90.0 kg at screening. BMI (kg/m^2) = Weight(kg) / {Height(m)}^2
* Decides to participate voluntarily in the study after being fully informed of and understanding the study completely, and provides his written informed consent prior to screening procedure.
* Determined eligible for this study in the opinion of the investigator based on the results of vital signs, physical examination, 12-lead electrocardiogram, clinical laboratory tests, and medical interview.

Exclusion Criteria:

* Has a history or current evidence of clinically significant disorder of hepatic, renal, nervous, respiratory, endocrine, hemato-oncologic, cardiovascular, urinary, and/or psychiatric system.
* Has a history or current evidence of gastrointestinal disease that may affect the safety and Pharmacokinetics assessment of investigational product(IP) or a history of gastrointestinal surgery (except for simple appendectomy or herniotomy).
* Has rheumatoid arthritis or has a history.
* Has symptomatic herpes simplex or herpes zoster or has a history within 3 months prior to the scheduled first dose.
* Has live vaccine dose within 3 months prior to the scheduled first dose or expects to receive live vaccine during the clinical trial period.
* Has a history or current evidence of clinically significant hypersensitivity to drugs containing any ingredient of Janus kinase inhibitor and other drugs.
* Has a positive result on serology tests (for hepatitis B, hepatitis C and human immunodeficiency virus [HIV], syphilis) during screening test.
* Has abnormalities one or more of the following during screening test: AST [GOT] or ALT [GPT] > 1.5 X upper limit of normal (ULN), Creatinine > upper limit of normal (ULN), ANC < 2,000/uL, Hb < 12.5 g/dL, Platelet < 150,000/uL, QTc interval at 12-lead electrocardiogram > 450 msec
* Systolic blood pressure (SBP) < 90 mmHg or > 140 mmHg, diastolic blood pressure (DBP) < 50 mmHg or > 95 mm Hg, or pulse rate (PR) < 45 beats/ min or > 100 beats/min on vital signs measured in sitting position after taking a rest for at least 5 minutes during screening test.
* Has a history of drug abuse or has a positive response to drug abuse on urine drug screening test.
* Has taken any prescription drugs or herbal medicine within 2 weeks prior to the expected date of first dose, or any over-the-counter (OTC) drug, health functional food or vitamin preparation within 1 week prior to the scheduled first dose (However, can participate in the study if otherwise eligible in the judgment of the investigator) or is expected to take such medication during the study.
* Has participated in any other clinical study, etc. and received IPs within 6 months prior to the scheduled first dose.
* Has donated whole blood within 2 months prior to the scheduled first dose, or has donated blood components or received transfusion within a month prior to the scheduled first dose.
* Has a history of excessive smoking (> 10 cigarettes/day) within 3 months prior to the scheduled first dose or confirmed as positive for cotinine on urine drug screening test.
* Excessive caffeine intake (> 5 units/day) or continued use of alcohol (> 21 units/week, 1 unit = 10 g of pure alcohol).
* Unable to stop drinking within 24 hrs prior to the scheduled first dose to post study visit.
* Unable to avoid caffeine-containing foods (e.g., coffee, tea [black tea, green tea, etc.], soda, coffee-flavored milk, and nutritive tonic drink, etc.) and foods containing grapefruit during each period from 24 hrs before hospitalization to discharge.
* Unable to use a medically acceptable contraceptive method stated below and does not agree not to donate sperm from the scheduled first dose to 90 days after the last dose.

  1. Use of intrauterine device with a proven birth control failure rate by the spouse (or partner)
  2. Simultaneous use of (male or female) barrier method and spermicide
  3. Surgical sterilization of the subject or his partner (e.g., vasectomy, salpingectomy, tubal ligation, or hysterectomy)
* Determined ineligible for study participation by the investigator for other reasons.

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-08-13 (Actual); Primary Completion 2022-02-24 (Estimated); Study Completion 2022-02-24 (Estimated)

PRIMARY OUTCOMES:
Cmax of IN-A002(IN-115314) | up to 72 hours
AUClast of IN-A002(IN-115314) | up to 72 hours

SECONDARY OUTCOMES:
AUCinf of IN-A002(IN-115314) | up to 72 hours
Tmax of IN-A002(IN-115314) | up to 72 hours
t1/2 of IN-A002(IN-115314) | up to 72 hours
λz of IN-A002(IN-115314) | up to 72 hours
CL/F of IN-A002(IN-115314) | up to 72 hours
Vd/F of IN-A002(IN-115314) | up to 72 hours
Cmax of IN-116118(primary metabolite of IN-A002(IN-115314)) | up to 72 hours
AUClast of IN-116118(primary metabolite of IN-A002(IN-115314)) | up to 72 hours
AUCinf of IN-116118(primary metabolite of IN-A002(IN-115314)) | up to 72 hours
Tmax of IN-116118(primary metabolite of IN-A002(IN-115314)) | up to 72 hours
t1/2 of IN-116118(primary metabolite of IN-A002(IN-115314)) | up to 72 hours
λz of IN-116118(primary metabolite of IN-A002(IN-115314)) | up to 72 hours
Metabolite ratio of IN-116118(primary metabolite of IN-A002(IN-115314)) | up to 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: In-Jin Jang, MD, PhD, Principal Investigator — Seoul National University Hospital, Dept. of Clinical Pharmacology
Locations (1):
- Seoul National University Hospital, Dept. of Clinical Pharmacology, Seoul, South Korea